CLINICAL TRIAL: NCT06735170
Title: Tuberoplasty Versus Balloon Spacer in Treatment of Rotator Cuff Tears
Brief Title: Tuberoplasty Versus Balloon Spacer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ORTHOSURG-2024-33151
Record Dates: First submitted 2024-12-03; First posted 2024-12-16 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Rotator Cuff Tears
Keywords: rotator cuff tear; shoulder surgery; tuberoplasty; subacromial balloon spacer
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Intervention Model Description: two armed study with each arm receiving one of two interventions: biologic tuberoplasty procedure or subacromial balloon spacer
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- biologic tuberoplasty group (Experimental): massive irreparable rotator cuff tear involving the supraspinatus and infraspinatus, no involvement of the subscapularis, centered humeral head on X-Ray examination, and a primary complaint of pain, randomized to biologic tuberoplasty surgery.
  Interventions: Procedure: biologic tuberoplasty
- subacromial balloon spacer group (Experimental): massive irreparable rotator cuff tear involving the supraspinatus and infraspinatus, no involvement of the subscapularis, centered humeral head on X-Ray examination, and a primary complaint of pain, randomized to subacromial balloon spacer.
  Interventions: Procedure: subacromial balloon spacer

INTERVENTIONS:
Procedure: biologic tuberoplasty — a surgical procedure during which an a cellular dermal allograft is attached to the greater tuberosity to prevent bone-to-bone contact between the greater tuberosity and the acromion with the goal of decreasing pain
  Arms: biologic tuberoplasty group
Procedure: subacromial balloon spacer — a biodegradable balloon is inserted into the subacromial space of the shoulder to increase teh distance between the greater tuberosity and the acromion to reduce pain
  Arms: subacromial balloon spacer group

SUMMARY:
The purpose of this study is to examine bone-to-bone contact between the tuberosity as compared to a subacromial balloon spacer procedure. Using biplanar fluoroscopy to determine the three-dimensional (3D) motion of the shoulder compared pre-procedure to post-procedure, the investigators will be able to assess 1) the bone-to-bone contact of the tuberosity and acromion in the setting of a massive posterior superior rotator cuff tear 2) if the placement of a dermal allograft over the tuberosity does indeed decrease bone contact and 3) if the placement of a subacromial balloon spacer decreases bone-to-bone contact. Doing so will allow assessment of the relative contribution of the implant for arm elevation versus potential compensatory motion of increased scapulothoracic motion. The investigators will also be able to correlate this to patient-reported outcomes of pain and shoulder function.

ELIGIBILITY:
Inclusion Criteria:

* Massive irreparable rotator cuff tear involving the supraspinatus and infraspinatus.
* No involvement of the subscapularis.
* Centered humeral head on X-ray examination.
* Primary complaint of pain.
* History of prior surgery, including failed rotator cuff repair.

Exclusion Criteria:

* Involvement of the subscapularis.
* Acromiohumeral distance less than 7 mm on upright anterior-posterior (AP) radiograph.
* Rotator cuff deemed repairable at the time of surgery.
* Patients younger than 65 years due to FDA clearance of the subacromial balloon spacer only for patients over 65

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2026-11-26 (Estimated); Study Completion 2026-11-26 (Estimated)

PRIMARY OUTCOMES:
change in bone-to-bone contact between tuberosity and acromion | presurgery, 6 months postop, 12 months postop
  degree of change in bone-to-bone contact between tuberosity and acromion as assessed using biplanar fluoroscopy
shoulder range of motion | presurgery, 1 week, 6 weeks, 3 months, 6 months, and 12 months postoperatively
  quantitative measurement in degrees with a goniometer of shoulder motion in forward elevation, abduction, external rotation, and internal rotation
single assessment numerical evaluation (SANE) of the shoulder | presurgery, 1 week, 6 weeks, 3 months, 6 months, and 12 months postoperatively
  a validated tool providing a numerical score from 0-100 that assess shoulder function as subjectively reported by the subject. A higher score indicates superior shoulder function.
American shoulder and elbow surgeons (ASES) score | presurgery, 1 week, 6 weeks, 3 months, 6 months, and 12 months postoperatively
  a validated survey with possible scores from 0-100 that assesses shoulder function as reported by the subject. A higher score indicates superior shoulder function.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Rao, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States